CLINICAL TRIAL: NCT07063472
Title: Effect of Kinesio Taping Versus Tele-Pilates Intervention on Pre-menstrual Syndrome
Brief Title: Kinesio Taping vs Tele-Pilates for PMS
Acronym: premensterual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Aly Elbandrawy, Professor of Physical Therapy for Women's Health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SREC SUE (1)325
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Premenstrual Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tele-Pilates (Experimental): The TP program included warm-up, main session, and cool-down phases. The session started with warm-up exercises in the form of breathing, spinal twist, cat stretch, arm circles, and abdominal stretching. Each exercise was performed for five repetitions, with each repetition held for 10-15 seconds and followed by a 5-second rest period. The warm-up phase lasted a total of 10 minutes.
  Tele-Pilates was supervised by a Pilates professional trainer. Participants engaged in mat-based Pilates exercises. These exercises included roll-up, bug leg, crock leg lying, prone single leg kick, bug roll, knee/lumbar roll, and prone attitude rotation. There was a 20-second rest in between the exercises. Each exercise was 3¬-5 reps, 10-¬15 sec hold, 5 secs rest. . The Pilates exercise protocol lasted for 8 weeks, with two sessions per week (totaling 16 sessions), each lasting 30 minutes. The session ended with 10-minute cool-down that involved relaxation exercises and stretching.
  Interventions: Behavioral: Tele- pilates
- Kinesio Tape (Other): Kinesio taping application for the KT group The participant sat upright in a chair, and a piece of kinesiology tape (5 × 5 cm, 3NS, Korea) was used to measure the distance from just above the anus to the upper border of the pelvis. This measured length was then divided by eight, and the tape was cut accordingly. One end of the tape was anchored on the ulnar bone just above the inguinal region. With 25% stretch, the tape was applied diagonally upward and outward, following the contour of the iliac crest over the ilium. The second end was secured to overlap the base of the initial tape. A second strip was applied in a similar manner in the opposite direction over the ilium. KT was applied for over eight weeks, with the tape changed every three days
  Interventions: Device: Kinesio taping application for the KT group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Tele- pilates — Tele-Pilates for (TP) group The TP program included warm-up, main session, and cool-down phases. The session started with warm-up exercises in the form of breathing, spinal twist, cat stretch, arm circles, and abdominal stretching. Each exercise was performed for five repetitions, with each repetition held for 10-15 seconds and followed by a 5-second rest period. The warm-up phase lasted a total of 10 minutes.
  Tele-Pilates was supervised by a Pilates professional trainer. Participants engaged in mat-based Pilates exercises. These exercises included roll-up, bug leg, crock leg lying, prone single leg kick, bug roll, knee/lumbar roll, and prone attitude rotation.The session ended with 10-minute cool-down that involved relaxation exercises and stretching.
  Arms: Tele-Pilates
Device: Kinesio taping application for the KT group — Kinesio taping application for the KT group The participant sat upright in a chair, and a piece of kinesiology tape (5 × 5 cm, 3NS, Korea) was used to measure the distance from just above the anus to the upper border of the pelvis. This measured length was then divided by eight, and the tape was cut accordingly. One end of the tape was anchored on the ulnar bone just above the inguinal region. With 25% stretch, the tape was applied diagonally upward and outward, following the contour of the iliac crest over the ilium. The second end was secured to overlap the base of the initial tape. A second strip was applied in a similar manner in the opposite direction over the ilium. KT was applied for over eight weeks, with the tape changed every three days
  Arms: Kinesio Tape

SUMMARY:
Premenstrual Syndrome (PMS) has a wide variety of signs and symptoms, including physical, psychological, and behavioral symptoms severe enough to disrupt daily activities. Objective: The study aimed to compare the effectiveness of a Tele-Pilates intervention and Kinesio Taping in managing symptoms of premenstrual syndrome (PMS).

DETAILED DESCRIPTION:
Ninety female participants aged 18 to 25 diagnosed with PMS were randomly assigned to one of three groups: the Kinesio Taping group (KT), the Tele-Pilates Exercise group (TP), or the Control group (CG). The KT group received taping intervention for eight weeks, the TP group engaged in an eight-week Tele-Pilates exercise program, while the CG maintained their usual routines without intervention. The Premenstrual Syndrome Questionnaire (PMSQ) was used to evaluate a range of PMS symptoms, including anxiety (PMS-A), depression (PMS-D), cravings (PMS-C), hyperhydration (PMS-H), other associated symptoms, and two menstruation-related symptoms: cramps and backache

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants had a regular menstrual cycle lasting 28 to 31 days for at least the previous three months, a visual analog scale (VAS) pain score of 4.0 or higher, and a normal body mass index (BMI)

Exclusion Criteria:

* Pelvic inflammatory disease or endometriosis
* The use of analgesics or oral contraceptives during the study period

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — For a study on Premenstrual Syndrome (PMS), eligibility should typically be limited to participants assigned female at birth who currently menstruate
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The Premenstrual Syndrome Questionnaire (PMSQ) | The participants answered the questionnaire items before the study course and after 8 weeks.
  The Premenstrual Syndrome Questionnaire (PMSQ) is a validated and reliable evaluation method for assessing PMS symptoms. It comprises five subscales: PMS-anxiety (PMS-A), PMS-depression (PMS-D), PMS-craving (PMS-C), PMS-hyperhydration (PMS-H), and a subscale for other associated symptoms. Additionally, the assessment includes two symptoms frequently reported during the initial two days of menstruation-cramps and backache. The PMS-A subscale addresses affective symptoms such as anxiety, irritability, mood swings, and nervous tension. PMS-D encompasses depressive symptoms, including depression, crying, forgetfulness, confusion, and insomnia. PMS-C evaluates somatic and behavioral symptoms such as increased appetite, headaches, fatigue, dizziness or fainting, and palpitations. PMS-H focuses on fluid retention, weight gain, breast tenderness, and abdominal bloating. The Other symptoms subscale covers a ra. The total PMSQ score ranges from 1 to 84, with higher scores indicating more severe

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Osthman O Doaa Osman, Assistant Professor, Study Director — Cairo University; Asmaa M. Elbandrawy, Professor, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy Outpatient Clinics, Alsalam University, Cairo, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: fficial website of the Kinesio Taping Association, offering clinical resources and background on the Kinesio Taping technique used in this study. — https://kinesiotaping.com/